CLINICAL TRIAL: NCT06948110
Title: Deciphering the Genetic Architecture of Autoimmune Diseases
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002412; 002412-HG
Record Dates: First submitted 2025-04-25; First posted 2025-04-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-04-23

CONDITIONS: Autoimmune Diseases
Keywords: Systemic Lupus Erythematosus
MeSH Terms: conditions — Autoimmune Diseases; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Affected: Person with an autoimmune disease

SUMMARY:
Background:

Autoimmune diseases can be caused by genes people inherit from their parents. The gene changes that cause these diseases have been well studied in people with European and Asian ancestors. But some diseases behave differently in people who are native to North and South America. Researchers want to know more about the gene changes and other factors that may cause autoimmune diseases among these people. This project will be based in Peru.

Objective:

To study how gene changes can lead to autoimmune diseases in people native to Peru.

Eligibility:

People aged 18 years and older with an autoimmune disease. These may include systemic lupus erythematosus; Sjogren disease; scleroderma; rheumatoid arthritis; seronegative spondylo-arthropathies; and systemic vasculitis. Family members and healthy volunteers are also needed.

Design:

Participants will have 2 clinic visits; these will be 2 weeks apart. The clinics will be in Lima, Iquitos, and other sites in Peru.

Visit 1: Participants will have a physical exam. They will answer questions about their health risks and habits. They will provide blood and urine samples.

Visit 2: Participants will provide a second blood sample and a stool sample. They will talk about the results of their first clinical exam with researchers.

The cost of travel to and from the clinics will be provided. Participants will get $30 per visit and a snack.

DETAILED DESCRIPTION:
SUMMARY:

The goal of this proposal is to investigate the genomic origins of heterogeneity in both risk and specific phenotype of autoimmune diseases, with a particular emphasis on understanding and addressing the health disparities of these diseases. Autoimmune diseases, especially Systemic Lupus Erythematosus (SLE), manifest at an earlier age and have worse clinical outcomes in individuals of non-European ancestry. Likewise, immunological genetic variants show a differential evolution based on geographical pathogenic pressure; almost 13 percent of loci for SLE, not including human leukocyte antigens (HLA), show signs of natural selection. Therefore, investigating the genomics of autoimmunity globally and in non-European populations is crucial to understanding these observations.

The prevalence of autoimmune diseases in Peru is difficult to estimate, since diagnoses require serologies that are not accessible, but it is estimated that there is a large proportion of undiagnosed or untreated cases in the country. Some studies conducted in Latin America and the United States report that the mestizo population presents SLE at an earlier age, with more systemic involvement than European populations. It is necessary to recognize that there is a significant gap in genomic studies conducted in the field of autoimmune diseases, revealing a serious underrepresentation in the indigenous populations of North and South America. In response to this critical need, collaborations have been established between physicians in different areas of Peru and Latin America to study the genomic architecture of autoimmunity in indigenous people in South America, carrying out cutting-edge genomic studies in this under-explored and high-risk population and evaluating population-specific genetic variants that may contribute to the identification of causal genes. including coding or structural changes. We propose to carry out state-of-the-art genomic studies in populations from different areas of Peru (Amazon, Andes, Coast) to describe the genomic architecture in this previously unstudied population.

General Objective:

The general objective of this project is to use genomic strategies to evaluate the molecular basis of human autoimmune diseases, representative of Peruvian populations. Diversification in genomic studies is necessary to reach personalized medicine and collaboration with community leaders and local researchers will ensure community participation and individual engagement, as well as training and education activities.

Specific Objectives:

Specific objective 1: To identify genetic markers associated with genetic risk of autoimmune diseases in the Indigenous population of Peru.

Specific objective 2: To evaluate the integrative multiomics (genomics, epigenomics and exposome) of the environmental context associated with autoimmunity in Peru.

Specific Objective 3: To characterize the microbiome in patients with autoimmunity in Peru.

Primary Endpoint:

Successful recruitment and whole-genome sequencing of at least 20 multiplex families with high familial autoimmunity burden, enabling identification and preliminary annotation of rare or novel genetic variants potentially linked to autoimmune disease susceptibility.

ELIGIBILITY:
* INCLUSION CRITERIA:

Any person who meets the criteria for inclusion in the study will be considered and must have the patient's signed informed consent for participation.

Autoimmune Disease Diagnosis:

Cases:

* Patients diagnosed with SLE, Sjogren's disease, scleroderma, rheumatoid arthritis, seronegative spondyloarthropathies, and systemic vasculitis, as defined by the American College of Rheumatology classification criteria.
* Over 18 years old

Controls:

* Family members of identified cases, and unrelated individuals. The controls would be from the same community as the patients and families studied, and of the same age and gender. Screening for autoimmune diseases and allergic diseases will be performed.
* Over 18 years old

EXCLUSION CRITERIA:

-People diagnosed with a chronic viral disease: HIV, hepatitis C or HTLV-1.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1) patients with suspected monogenic disorders of germinal origin and/or early-onset systemic lupus erythematosus; 2) families with multiple individuals with systemic lupus erythematosus and a history of consanguinity; 3) belonging to an isolated population; and 4) families with high autoimmunity penetrance.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2030-04-22 (Estimated); Study Completion 2030-04-22 (Estimated)

PRIMARY OUTCOMES:
whole-genome sequencing | Ongoing
  Successful recruitment and whole-genome sequencing of at least 20 multiplex families with high familial autoimmunity burden, enabling identification and preliminary annotation of rare or novel genetic variants potentially linked to autoimmune disease susceptibility.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina M Lanata, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States
- Amazon Rainforest, Lima, Peru

IPD SHARING:
Plan to Share IPD: No